CLINICAL TRIAL: NCT02641015
Title: A Retrospective Observational Study to Assess the Clinical Management and Outcomes of Hospitalised Patients With Complicated Urinary Tract Infection in Countries With High Prevalence of Multidrug Resistant Gram-negative Bacteria.
Brief Title: Study to Assess Management and Outcomes of Hospitalised Patients With Complicated UTI (RESCUING)
Acronym: RESCUING
Status: Completed | Type: Observational
Sponsor: Institut d'Investigació Biomèdica de Bellvitge (Other)
Collaborators: Tel Aviv University (Other); AiCuris Anti-infective Cures AG (Industry); University of Bristol (Other); UMC Utrecht (Other)
Responsible Party: Principal Investigator, Miquel Pujol, PhD, Institut d'Investigació Biomèdica de Bellvitge
Other Study IDs: PR 223/15
Record Dates: First submitted 2015-12-23; First posted 2015-12-29 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Urinary Tract Infections; Bacterial Resistance
Keywords: UTI
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
A retrospective observational study to assess the clinical management and outcomes of hospitalised patients with complicated urinary tract infection in countries with high prevalence of multidrug resistant gram-negative bacteria (COMBACTE-MAGNET,WP5)

DETAILED DESCRIPTION:
Bacterial resistance to antimicrobial drugs is a major public health problem. Of greatest concern is the rapid emergence and dissemination of resistance to third generation cephalosporins in Enterobacteriaceae, especially Escherichia coli and Klebsiella pneumoniae. This is frequently seen in association with resistance to other classes of antibiotics leading to a multidrug resistance (MDR) profile. These MDR isolates are often involved in complicated urinary tract infection (cUTI), and are associated with poor clinical outcomes. In addition, in the last decade there has been an emergence of carbapenemase-producing Enterobacteriaceae, which are also resistant to other antibiotics than carbapenems, leaving few therapeutic options.

The overall aim of this study is to provide information about the epidemiology, clinical management and outcome of patients hospitalised with cUTI, including pyelonephritis. To achieve this aim, the investigators will perform a multicentre retrospective observational study in patients with hospitalised cUTI. The study will be conducted in several European countries plus Israel, which have a high prevalence of MDR Gram-negative bacteria (GNB), including Pseudomonas aeruginosa. The study will seek to identify possible modifiable risk factors for treatment failure, especially those related to antibiotic therapy.

On completion of this study, the investigators will develop a better understanding of the clinical management of hospitalised patients with cUTI due to MDR GNB in European countries. The investigators will identify the modifiable risk factors for treatment failure. This information will be used to inform better clinical and antibiotic management of cUTI to improve patient outcomes. The study will also be used in the development of hypothesis for future randomised controlled trials in cUTI with new antibiotics. Dissemination of results will take place through peer-reviewed publications and conference presentations.

ELIGIBILITY:
Inclusion Criteria:

Patients with UTI and at least one of the following underlying conditions:

* Indwelling urinary catheter
* Urinary retention (at least 100ml of residual urine after voiding)
* Neurogenic bladder
* Obstructive uropathy (e.g. nephrolithiasis, fibrosis)
* Renal impairment caused by intrinsic renal disease: Estimated glomerular filtration rate (eGFR) <60 mL/min
* Renal transplantation
* Urinary tract modifications, such as an ileal loop or pouch
* Pyelonephritis and normal urinary tract anatomy

and at least one of the following signs or symptoms:

* Chills or rigors associated with fever or hypothermia (temperature greater than 38ºC or below 36ºC)
* Flank pain (pyelonephritis) or pelvic pain (cUTI)
* Dysuria, urinary frequency, or urinary urgency
* Costo-vertebral angle tenderness on physical examination
* UTI-related altered mental state

and at least one of the following microbiological results:

* Urine culture with at least 105 CFU/mL or greater of a uropathogen (no more than 2 species)
* At least one blood culture growing possible uropathogens (no more than 2 species) with no other evident site of infection

Exclusion Criteria:

* Patients less than 18 years of age
* Prostatitis
* Polymicrobial infections that include Candida spp.
* Polymicrobial infections that include more than 2 bacterial species
* cUTI with Candida spp. as sole uropathogen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalised patients from 1st January 2013 to the 31st December 2014. Diagnosis of cUTI as the primary cause of hospitalisation and patients hospitalised for another reason but who developed cUTI during their hospitalisation. Patients will be identified by searching for any of the following ICD-9 CM or ICD-10 CM codes at discharge on the hospital administration system: ICD-9 CM Codes: 590.1, 590.10, 590.11, 590.2, 590.8, 590.80, 590.9, 595.0, 595.89, 595.9, 99.0 ICD-10 CM Codes: N10, N12, N13.6, N15.1, N15.9, N30.0, N30.8, N30.9, N39.0
Sampling Method: Non-Probability Sample
Enrollment: 1028 (Actual)
Dates: Start 2015-12; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Treatment Failure | 30 days
  Treatment failure will be assessed as number of participants with evidence of treatment failure or mortality within 30 days from initial cUTI diagnosis

SECONDARY OUTCOMES:
Time to clinical response | 30 days
  Time to clinical response (in days), since initiation of antibiotic treatment
Time to urological intervention for source control | 30 days
  Time to urological intervention for source control (in days) since initial cUTI diagnosis
Time to death | 30 days
  Time to death (in days) since original cUTI diagnosis
Duration of antibiotic therapy | 30 days
  Duration of antibiotic therapy (in days)
Length of hospital stay | 30 days
  Length of hospital stay (in days)
Hospital mortality | 30 days
  Hospital mortality during admission
All cause mortality within 30 days of the original cUTI diagnosis | 30 days
  All cause mortality within 30 days of the original cUTI diagnosis
All cause of mortality for two months after hospital discharge | 60 days
  All cause of mortality for two months after hospital discharge
Cost per case of cUTI | 30 days
  Cost per case of cUTI
Readmissions to the hospital within 60 days of hospital discharge | 60 days
  Readmissions to the hospital within 60 days of hospital discharge
Adverse events related to antibiotic treatment including: moderate or severe allergic reactions, severe renal impairment, Clostridium difficile infection | 30 days
  Adverse events related to antibiotic treatment including: moderate or severe allergic reactions, severe renal impairment, Clostridium difficile infection

CONTACTS AND LOCATIONS:
Overall Officials: Dora Tancheva, Mrs, Principal Investigator — Emergency Hospital Pirogov, Sofia, Bulgaria; Rossitza Vatcheva-Dobrevska, Prof, Principal Investigator — University Hospital Queen Joanna, Sofia, Bulgaria; Sotirios Tsiodras, Prof, Principal Investigator — Attikon University Hospital, Athens, Greece; Emmanuel Roilides, Prof, Principal Investigator — Hippokration Hospital, Thessaloniki, Greece; Istvan Vakonyi, MD, Principal Investigator — Kenezy University Hospital,Debrecen, Hungary; Aniko Farkas, MD, Principal Investigator — Szabolcs-Szatmár-Bereg Megyei Kórházak és Egyetemi Oktatókórház (SZSZBMK). Nyíregyháza, Hungary; Leonard Leibovici, Prof, Principal Investigator — Beilinson Hospital, Rabin Medical Center. Petah-TiqvaI, Israel; Mical Paul, Prof, Principal Investigator — Rambam Health Care Campus. Haifa, Israel; Yehuda Carmeli, Prof, Principal Investigator — Tel Aviv Medical Center, Tel Aviv. Israel; Emanuele Durante Mangoni, Prof, Principal Investigator — AORN dei Colli Monaldi. Napoli, Italy; Erica Franceschini, MD, Principal Investigator — Azienda ospedaliero-universitaria policlinico di modena, Modena, Italy; Nicola Petrosillo, MD, Principal Investigator — National Institute for Infectious Diseases L. Spallanzani, IRCCS, Rome, Italy; Andrei Ursache, MD, Principal Investigator — "Spitalul Clinic de Urgenta Bucuresti. Popular unoficial name ""Floreasca "" Hospital", Bucharest, Romania; Judit BodnÃ¡r, MD, Principal Investigator — Soproni Erzsébet Oktató Kórház és Rehabilitációs Intézet, Sopron, Hungary; Yehuda Carmeli, Prof, Principal Investigator — Tel Aviv Medical Center, Tel Aviv, Israel; Andrei Vata, MD, Principal Investigator — Infectious Diseases Hospital Sfanta Parascheva Iasi, Iasi, Romania; Adriana Hristea, MD, Principal Investigator — National Institute for Infectious Diseases Prof Dr Matei Bals, Bucharest, Romania; Jesus Rodriguez-Bano, Prof, Principal Investigator — Hospital Universitario Virgen Macarena, Seville, Spain; Julia Origüen, MD, Principal Investigator — Hospital Universitario 12 de Octubre, Madrid, Spain; Arzu Yetkin, MD, Principal Investigator — Ankara Numune Egitim ve ArastÄrma Hastanesi, Ankara, Turkey; Nese Saltoglu, Prof, Principal Investigator — Istanbul University Cerrahpasa Medical School, Istambul, Turkey; Miquel Pujol, MD, Principal Investigator — Hospital Universitari de Bellvitge, Barcelona, Spain
Locations (21):
- Bulgaria (2):
  - Emergency Hospital Pirogov, Sofia
  - University Hospital Queen Joanna, Sofia
- Greece (2):
  - Attikon University Hospital, Athens
  - Hippokration Hospital, Thessaloniki
- Hungary (3):
  - Kenezy University Hospital, Debrecen
  - Szabolcs-Szatmár-Bereg Megyei Kórházak és Egyetemi Oktatókórház (SZSZBMK), Nyíregyháza
  - Soproni Erzsébet Oktató Kórház és Rehabilitációs Intézet, Sopron
- Israel (3):
  - Rambam Health Care Campus, Haifa
  - Beilinson Hospital, Rabin Medical Center, Petah Tikva
  - Tel Aviv Medical Center, Tel Aviv
- Italy (3):
  - Azienda Ospedaliero-Universitaria Policlinico Di Modena, Modena
  - AORN dei Colli Monaldi, Napoli
  - National Institute for Infectious Diseases L. Spallanzani, IRCCS, Rome
- Romania (3):
  - "Spitalul Clinic de Urgenta Bucuresti. Popular unoficial name ""Floreasca "" Hospital", Bucharest
  - National Institute for Infectious Diseases Prof Dr Matei Bals, Bucharest
  - Infectious Diseases Hospital Sfanta Parascheva Iasi, Iași
- Spain (3):
  - Hospital Universitari de Bellvitge, L'Hospitalet Del Llobregat, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Virgen Macarena, Seville
- Turkey (Türkiye) (2):
  - Ankara Numune Egitim ve ArastÄ±rma Hastanesi, Ankara
  - Istanbul University Cerrahpasa Medical School, Istanbul

REFERENCES:
- [Background] Morrissey I, Hackel M, Badal R, Bouchillon S, Hawser S, Biedenbach D. A Review of Ten Years of the Study for Monitoring Antimicrobial Resistance Trends (SMART) from 2002 to 2011. Pharmaceuticals (Basel). 2013 Nov 1;6(11):1335-46. doi: 10.3390/ph6111335. PMID 24287460
- [Background] Hoban DJ, Lascols C, Nicolle LE, Badal R, Bouchillon S, Hackel M, Hawser S. Antimicrobial susceptibility of Enterobacteriaceae, including molecular characterization of extended-spectrum beta-lactamase-producing species, in urinary tract isolates from hospitalized patients in North America and Europe: results from the SMART study 2009-2010. Diagn Microbiol Infect Dis. 2012 Sep;74(1):62-7. doi: 10.1016/j.diagmicrobio.2012.05.024. Epub 2012 Jul 2. PMID 22763019
- [Background] Yang YS, Ku CH, Lin JC, Shang ST, Chiu CH, Yeh KM, Lin CC, Chang FY. Impact of Extended-spectrum beta-lactamase-producing Escherichia coli and Klebsiella pneumoniae on the outcome of community-onset bacteremic urinary tract infections. J Microbiol Immunol Infect. 2010 Jun;43(3):194-9. doi: 10.1016/S1684-1182(10)60031-X. PMID 21291846
- [Background] Ha YE, Kang CI, Cha MK, Park SY, Wi YM, Chung DR, Peck KR, Lee NY, Song JH. Epidemiology and clinical outcomes of bloodstream infections caused by extended-spectrum beta-lactamase-producing Escherichia coli in patients with cancer. Int J Antimicrob Agents. 2013 Nov;42(5):403-9. doi: 10.1016/j.ijantimicag.2013.07.018. Epub 2013 Sep 7. PMID 24071027
- [Background] Trecarichi EM, Tumbarello M. Antimicrobial-resistant Gram-negative bacteria in febrile neutropenic patients with cancer: current epidemiology and clinical impact. Curr Opin Infect Dis. 2014 Apr;27(2):200-10. doi: 10.1097/QCO.0000000000000038. PMID 24573013
- [Background] Kumar A, Ellis P, Arabi Y, Roberts D, Light B, Parrillo JE, Dodek P, Wood G, Kumar A, Simon D, Peters C, Ahsan M, Chateau D; Cooperative Antimicrobial Therapy of Septic Shock Database Research Group. Initiation of inappropriate antimicrobial therapy results in a fivefold reduction of survival in human septic shock. Chest. 2009 Nov;136(5):1237-1248. doi: 10.1378/chest.09-0087. Epub 2009 Aug 20. PMID 19696123
- [Background] Spoorenberg V, Hulscher ME, Akkermans RP, Prins JM, Geerlings SE. Appropriate antibiotic use for patients with urinary tract infections reduces length of hospital stay. Clin Infect Dis. 2014 Jan;58(2):164-9. doi: 10.1093/cid/cit688. Epub 2013 Oct 24. PMID 24158412
- [Background] Levison ME, Kaye D. Treatment of complicated urinary tract infections with an emphasis on drug-resistant gram-negative uropathogens. Curr Infect Dis Rep. 2013 Apr;15(2):109-15. doi: 10.1007/s11908-013-0315-7. PMID 23378123
- [Background] Nicolle LE. A practical guide to the management of complicated urinary tract infection. Drugs. 1997 Apr;53(4):583-92. doi: 10.2165/00003495-199753040-00004. PMID 9098661
- [Background] Foxman B. Epidemiology of urinary tract infections: incidence, morbidity, and economic costs. Am J Med. 2002 Jul 8;113 Suppl 1A:5S-13S. doi: 10.1016/s0002-9343(02)01054-9. PMID 12113866
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] Karnofsky DA, Burchenal JH: The clinical evaluation of chemotherapeutic agents in cancer. In Evaluation of chemotherapeutic agents. Edited by MacLeod CM. New York: Columbia University Press; 1949:191-205.
- [Background] Barber J, Thompson S. Multiple regression of cost data: use of generalised linear models. J Health Serv Res Policy. 2004 Oct;9(4):197-204. doi: 10.1258/1355819042250249. PMID 15509405
- [Background] Magiorakos AP, Srinivasan A, Carey RB, Carmeli Y, Falagas ME, Giske CG, Harbarth S, Hindler JF, Kahlmeter G, Olsson-Liljequist B, Paterson DL, Rice LB, Stelling J, Struelens MJ, Vatopoulos A, Weber JT, Monnet DL. Multidrug-resistant, extensively drug-resistant and pandrug-resistant bacteria: an international expert proposal for interim standard definitions for acquired resistance. Clin Microbiol Infect. 2012 Mar;18(3):268-81. doi: 10.1111/j.1469-0691.2011.03570.x. Epub 2011 Jul 27. PMID 21793988
- [Derived] Shaw E, Addy I, Stoddart M, Vank C, Grier S, Wiegand I, Leibovici L, Eliakim-Raz N, Vallejo-Torres L, Morris S, MacGowan A, Carratala J, Pujol M; COMBACTE-MAGNET Consortium. Retrospective observational study to assess the clinical management and outcomes of hospitalised patients with complicated urinary tract infection in countries with high prevalence of multidrug resistant Gram-negative bacteria (RESCUING). BMJ Open. 2016 Jul 29;6(7):e011500. doi: 10.1136/bmjopen-2016-011500. PMID 27473949
- See also: UK Five Year Antimicrobial Resistance Strategy 2013-2018, September 2013. — http://www.gov.uk/government/uploads/system/uploads/attachment_data/file/244058/20130902_UK_5_year_AMR_strategy.pdf
- See also: Complicated Urinary Tract Infections: Developing Drugs for Treatment. Guidance for Industry (2015). U.S. Department of Health and Human Services, Food and Drug Administration Center for Drug Evaluation and Research (CDER). — http://www.fda.gov/downloads/Drugs/Guidances/ucm070981.pdf
- See also: International Classification of Diseases ICD-9 Data. — http://icd9data.com/2015/volume1/580-629/default.htm
- See also: International Statistical Classification of diseases and related Health Problems 10th Revision. ICD-10. Version 2015. — http://apps.who.int/classifications/icd10/browse/2015/en
- See also: University of Maryland Medical Center. Urinary tract Infection — http://umm.edu/health/medical/reports/articles/urinary-tract-infection
- See also: Directive 95/46/EC of the European Parliament and of the Council of 24 October 1995 on the protection of individuals with regard to the processing of personal data and on the free movement of such data — http://eur-lex.europa.eu/legal-content/GA/ALL/?uri=OJ:L:1995:281:TOC